CLINICAL TRIAL: NCT05888506
Title: The Effects of Ketone Ester Supplementation on Nocturnal Blood Pressure in Middle-Aged and Older Adults
Brief Title: Ketone Ester Supplementation and Nocturnal Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Southern University (Other)
Collaborators: Auburn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H23223
Record Dates: First submitted 2023-04-05; First posted 2023-06-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases in Old Age; Aging; Cardiovascular Diseases; Sleep
Keywords: blood pressure; sleep; heart rate variability; ketone ester
MeSH Terms: conditions — Cardiovascular Diseases | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone Ester (Experimental): Participants will consume the supplement prior to bedtime. Nocturnal blood pressure, heart rate, and sleep characteristics will be assessed
  Interventions: Dietary Supplement: Ketone Ester
- Placebo Supplement (Placebo Comparator): Participants will consume the supplement prior to bedtime. Nocturnal blood pressure, heart rate, and sleep characteristics will be assessed
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Ester — Participants will consume the ketone ester beverage produced by KetoneAid prior to bedtime. Participants will consume 60 mL (30 grams ketones) of the ketone beverage.
  Arms: Ketone Ester
Dietary Supplement: Placebo — Participants will consume the placebo supplement prior to bedtime. The placebo supplement will be a ketone ester-free, taste and viscosity-matched, beverage produced by KetoneAid.
  Arms: Placebo Supplement

SUMMARY:
Cardiovascular disease (CVD) is the number one cause of death globally and high blood pressure (i.e., hypertension) is the leading modifiable risk factor for CVD and all-cause mortality. Advancing age is the primary risk factor for hypertension and CVD. Moreover, compared to younger adults, older adults exhibit reduced nocturnal dipping of blood pressure resulting in elevated nighttime blood pressure values, which are a better predictor of cardiovascular outcomes than daytime blood pressure. Intriguingly, recently published rodent data suggests that ketone supplementation protects against hypertension, blood vessel dysfunction, and kidney injury. Whether ketone supplementation provides vascular health benefits in humans remains to be determined. Therefore, the investigations seek to conduct an acute ketone supplementation study to determine whether ketone supplementation may restore a more healthy nighttime blood pressure phenotype in middle-aged and older adults. The investigations will also determine whether ketone supplementation influences nocturnal heart rate variability, a non-invasive of autonomic function that may be influenced by ketone supplementation in a manner that influences blood pressure.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death globally, killing one American approximately every 40 seconds. Among known risk factors, hypertension, or high blood pressure (BP), is the most important risk factor for the development of CVD. While sleeping, a healthy adult will experience a blood pressure dip of about 10% compared to resting values while awake. However, advancing age is associated with reduced blood pressure dipping, which is linked with an increased risk for CVD. Moreover, attenuated blood pressure dipping results in elevated nighttime blood pressure, which is in general a better predictor of cardiovascular outcomes than daytime blood pressure.

The autonomic nervous system plays a key role in blood pressure regulation and autonomic dysregulation is implicated in the pathophysiology of hypertension. Advancing age is associated with structural and function changes in the autonomic nervous system, which likely contribute, at least in part, to the marked elevation in the prevalence of hypertension and CVD that is observed in older adults. Heart rate variability (HRV) is an inexpensive and accessible index of autonomic function that is shown to decline rapidly form the second to fifth decades of life. Thus, strategies to improve nocturnal HRV may help to restore a more healthy nighttime blood pressure phenotype. However, this remains to be proven. Moreover, the link between aging, nocturnal HRV, and nighttime blood pressure is unclear.

Hypertension costs the United States between $131 and $198 billion dollars each year. Therefore, there exists a critical need to find ways to mitigate these negative health effects and costs to both the American public, and populations across the globe. Interestingly, there is a small but emerging body of evidence suggesting that ketone bodies may positively impact endothelial function and vascular health. In rodents, ketone supplementation prevents high-salt induced increase in blood pressure, blood vessel dysfunction, and kidney injury. However, there is a lack of data regarding whether ketone supplementation may provide similar cardiovascular health benefits in humans. Thus, in this first-of-kind placebo-controlled, randomized crossover design acute ketone supplementation study the investigations will evaluate the hypothesis that acute ketone supplementation will improve nocturnal blood pressure and HRV in middle-aged and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 50 years of age
* Body mass index (BMI) below 40 kg/m^2
* No alterations to use of prescription medication within the past 6 months

Exclusion Criteria:

* Alterations to use of prescription medication within the past 6 months
* Allergy to any of the ingredients in the ketone beverage
* Communication barriers

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Nocturnal blood pressure dipping | Night one of supplement ingestion (i.e., from time asleep to time awake for one night per condition)
  The investigations will use ambulatory blood pressure monitoring to characterize night-to-day blood pressure ratio

SECONDARY OUTCOMES:
Nighttime blood pressure | Night one of supplement ingestion (i.e., from time asleep to time awake for one night per condition)
  The investigations will use ambulatory blood pressure monitoring to characterize nighttime blood pressure (mmHg)
Nighttime heart rate variability | Night one of supplement ingestion (i.e., from time asleep to time awake for one night per condition)
  The investigators will use a single-lead electrocardiograph to characterize nocturnal heart rate variability (ms)
Objective sleep duration | Night one of supplement ingestion (i.e., from time asleep to time awake for one night per condition)
  Actigraph accelerometers will be used to quantify sleep duration
Objective sleep efficiency | Night one of supplement ingestion (i.e., from time asleep to time awake for one night per condition)
  Actigraph accelerometers will be used to quantify % of time in bed actually spent sleeping to calculate sleep efficiency
Subjective sleep quality | Night one of supplement ingestion (i.e., from time asleep to time awake for one night per condition)
  A single-item visual analogue sleep scale will be used to quantify subjective sleep quality (i.e., 0 to 100, with a higher score indicating better sleep)
Subjective sleep quality | Pre-intervention
  The investigators will use the Pittsburgh Sleep Quality Index (PSQI) to assess perceived sleep quality reflective of the one month period leading into the study. PSQI scores range from 0-21, with a higher score indicting worse sleep.
Pulse wave analysis | Pre-intervention
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA) The sampling site is the brachial artery (upper alarm instrumented with a cuff for oscillometric sphygmomanometer).
Pulse wave velocity | Pre-intervention
  The investigators will use the SphygmoCor XCEL system to assess pulse wave velocity (PWV). A high-fidelity strain-gauge transducer is used to obtain the pressure waveform at the carotid pulse. Distances from the carotid artery sampling site to the femoral artery (upper leg instrumented with a thigh cuff for oscillometric sphygmomanometry), and from the carotid artery to the suprasternal notch will be recorded. PWV will be expressed as m/s.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Grosicki, PhD, Principal Investigator — Georgia Southern University
Locations (1):
- Biodynamics and Human Performance Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fagard RH, Celis H, Thijs L, Staessen JA, Clement DL, De Buyzere ML, De Bacquer DA. Daytime and nighttime blood pressure as predictors of death and cause-specific cardiovascular events in hypertension. Hypertension. 2008 Jan;51(1):55-61. doi: 10.1161/HYPERTENSIONAHA.107.100727. Epub 2007 Nov 26. PMID 18039980
- [Background] Valensi P. Autonomic nervous system activity changes in patients with hypertension and overweight: role and therapeutic implications. Cardiovasc Diabetol. 2021 Aug 19;20(1):170. doi: 10.1186/s12933-021-01356-w. PMID 34412646
- [Background] Chakraborty S, Galla S, Cheng X, Yeo JY, Mell B, Singh V, Yeoh B, Saha P, Mathew AV, Vijay-Kumar M, Joe B. Salt-Responsive Metabolite, beta-Hydroxybutyrate, Attenuates Hypertension. Cell Rep. 2018 Oct 16;25(3):677-689.e4. doi: 10.1016/j.celrep.2018.09.058. PMID 30332647